CLINICAL TRIAL: NCT01654861
Title: Evaluation of the Safety and Efficacy of Standard Dose Gemcitabine Combined With High Dose Intravenous Vitamin C (HDIVC) Treatment for Patients With Metastatic Adenocarcinoma of the Pancreas.
Brief Title: Safety & Efficacy Study of Gemcitabine...With High Dose IV Vit. C (HDIVC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: recruiting or enrolling participants has halted prematurely and will not resume
Sponsor: Eastern Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERMC 11-11
Record Dates: First submitted 2012-07-13; First posted 2012-08-01 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-01

CONDITIONS: Metastatic Adenocarcinoma of the Pancreas
MeSH Terms: interventions — Gemcitabine; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HDIVC (Experimental): Gemcitabine (Gemzar), Intravenous and oral Ascorbic Acid (Vitamin C).
  Interventions: Drug: Gemcitabine, Intravenous and oral Ascorbic Acid (Vitamin C)

INTERVENTIONS:
Drug: Gemcitabine, Intravenous and oral Ascorbic Acid (Vitamin C) — Weeks 1,2,3: IV Gemcitabine 1000 mg / m² over 30 minutes followed by HDIVC 1.2 g / kg: 1.2 g/kg over 90 minutes for a dose ≤90 g and over 120 minutes for a dose >90g followed by 0.3 g / kg over 120 minutes; Week 4: no treatment.

SUMMARY:
* The combination of gemcitabine and HDIVC is safe and may favorably change the clinical course for an individual patient.
* The combination of gemcitabine and HDIVC is synergistic in anti-tumor effect as seen in preclinical models, where HDIVC creates a pro-oxidative effect that adds to the anti-tumor effect of gemcitabine.
* The combination of gemcitabine and HDIVC may improve Progression Free Survival (PFS).
* The dosage schema of 1.2 g /kg bolus infusion followed by lower dose of 0.3 g / kg infusion may create sustained elevation in Vitamin C plasma levels for increased cytotoxic effect.
* The addition of HDIVC & oral supplementation of Vitamin C to standard treatment with gemcitabine may improve quality of life for patients with comparison to prior to treatment start of this protocol.
* CA 19-9 and inflammatory markers may show trends for patients in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age
* Biopsy proven adenocarcinoma of the pancreas
* Evidence of metastatic disease
* Received at least 1 prior chemotherapy treatment regimen with disease progression
* May have had any prior chemotherapy regimen including any gemcitabine based regimen or FOLFIRINOX
* May have participated in a prior study protocol
* May have had prior treatment with HDIVC
* Anticipated survival of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status = 0,1, or 2
* The patient must have screening laboratory: ANC ≥ 1,500/mm3, Hemoglobin > 8g/dL, Platelets ≥ 100,000/mm3, Total Bilirubin < 1.5mg/dL, Creatinine ≤ 1.5mg/dL, Transaminases < 2.5 x upper limit of normal, Urine Uric Acid < 1.000 mg/d, Urine pH < 6, Urine microscopic negative for oxalates (if positive, reflex urinary oxalates < 60mg/d), PT INR ≤ 1.5, unless patient is on full dose warfarin
* Glucose-6-phosphate dehydrogenase deficiency (G6PD) normal status via blood test The fluorescent spot test is the simplest, most reliable, and most sensitive of the G6PD screening tests
* Willingness to undergo central line placement and able to manage care of the entry site safely
* Willingness to adhere to supplemental oral dose regimen of ascorbic acid 500mg taken twice daily
* All other nutritional supplements would be discontinued for the duration of the trial except for pancreatic enzymes and probiotics
* Patients must be able to take food orally or have a peg tube for feeding
* Able to give consent for protocol participation

Exclusion Criteria:

* Glucose-6-phosphate dehydrogenase deficiency (G6PD)
* Renal insufficiency : serum creatinine of > 1.5 mg /dl or evidence of oxalosis by urinalysis prior to enrollment and prior to each HDIVC infusion
* Documentation or report of history of kidney stones or urinary oxalosis.
* Co-morbid condition that would affect survival: congestive heart failure, unstable angina, myocardial infarction within 6 weeks of study, uncontrolled blood sugars of > 300 mg / dl, patients with known chronic active hepatitis or cirrhosis
* Currently active second malignancy
* Chronic hemodialysis
* Iron overload/ Hemochromatosis: Ferritin > 500 ng / ml
* Wilson's disease
* Pregnant or lactating female (pre- menopausal females will undergo pregnancy test prior to administration of protocol drugs throughout treatment cycles during this study)
* Aspirin use exceeding 81 mg per day
* Acetaminophen use exceeding 2 g per day
* Known brain metastasis
* Active tobacco smokers
* Treatment with the combination of HDIVC and gemcitabine previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eiko Klimant, MD, FACP, Principal Investigator — Eastern Regional Medical Center; Heather Wright, ND, FABNO, Principal Investigator — Eastern Regional Medical Center
Locations (1):
- Eastern Regional Medical Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HDIVC
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HDIVC
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 55 [52 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events as a Measure of Safety and Tolerability
Description: Adverse events, whether volunteered by the study subject, discovered by the investigators during questioning, or detected by physical examination, laboratory tests, or other means will be collected and recorded at each visit. Events will be recorded from the time the consent is signed until 4 weeks after the study protocol is discontinued. Subjects experiencing Grade 4 neutropenia, Grade ≥3 thrombocytopenia, or Grade 2 peripheral neuropathy who do not recover will have treatment protocol discontinued.
Time Frame: Weekly for up to 6 months.
Measure: Number; unit: participants
Arm/Group | HDIVC
Number analyzed (Participants) | 3
participants | 0

2. Secondary Outcome: Anti-Tumor Response
Description: CT and PET scans will be performed at baseline and then every two months. Target and Non-Target Lesions will be identified and recorded at baseline. When subsequent scans are performed, anti-tumor responses will be assessed using Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Every 2 months for up to 6 months.
Population: Data were not analyzed as the study was prematurely closed.
Arm/Group | HDIVC
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | HDIVC
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes